CLINICAL TRIAL: NCT03346499
Title: Adoptive Transfer of Haploidentical Natural Killer Cells and IL-2 in Human Immunodeficiency Virus (HIV)
Brief Title: Adoptive Transfer of Haploidentical Natural Killer Cells and IL-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1508M77601-2
Record Dates: First submitted 2017-10-24; First posted 2017-11-17 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: HIV
Keywords: HIV
MeSH Terms: interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NK cells and IL-2 (Experimental)
  Interventions: Biological: NK cells and IL-2

INTERVENTIONS:
Biological: NK cells and IL-2 — Natural Killer Cells

SUMMARY:
This is a pilot study of the infusion of haploidentical NK cells with IL-2 in 5 HIV+ individuals who are on stable ART with full HIV suppression.

DETAILED DESCRIPTION:
Potential subjects will be screened to determine eligibility. Immediately after consent and screening, an HLA-haploidentical donor will be identified and will complete eligibility screen and consent. At Day -7 the subject will undergo an inguinal lymph node biopsy and colonoscopy to obtain ileal and rectal biopsies. Blood samples will be obtained to measure chimerisms, plasma HIV RNA, and inflammatory cytokines. PBMCs will be obtained to sort into CD4 subsets and measure frequencies of HIV RNA and DNA. On Day -1, the donor will undergo apheresis and donor cells will be obtained and incubated overnight with IL-2. On Day 0 subjects will start aspirin and be infused with IL-2 activated NK cells. Subjects will receive 6 million units of IL-2 just after the infusion and they will be monitored on the Phase 1 Unit for 24 hours. Plasma will be obtained at 2 hrs, 4 hrs and the following morning and stored for measures of inflammatory markers. The subject will return to the outpatient clinic on days 2, 4, 6, 8, and 10 after the infusion for administration of 6 million units of IL-2 and to obtain plasma and PBMC for measures of inflammatory markers and changes to the virus reservoir. On day 14 the subject will stop taking ASA and blood will be obtained to measure frequencies of HIV RNA and DNA. On day 21 will have a lymph node biopsy and colonoscopy to obtain ileal and rectal tissues. The patient will then be followed until day 100 post NK cell infusion. Subjects will return every 2 weeks for a toxicity assessment, blood draws, and viral level testing. Study participation will end after day 100.

ELIGIBILITY:
Inclusion Criteria:

* ¥ Age-18-65

  * Stable ART for at least 12 months.
  * Screening plasma HIV RNA levels below level of quantification (<40 to <50 copies RNA/mL depending on the assay) for ≥ 6 months (a total of 3 measurements above the level of detection but < 500 copies/ml will be allowed if each detectable measure is separated by at least 1 year)
  * Screening CD4 count ≥500 cells/µl
  * Laboratory tests (CBCD, CMP, Mg, Phosphorus, PT/PTT, TSH/T4,) performed within 14 days of study enrollment. All laboratory results (unless otherwise specified) must be Grade 1 or normal based on the DAIDS Adverse Event Grading Scale (Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events v2.0)
  * Adequate kidney function defined by estimated GFR (CrCl) > 60 ml/min or ml/min/1.73 m2 (≤ grade 2 per DAIDS) and creatinine ≤ 1.5 x ULN
  * Adequate pulmonary function without any clinical signs or symptoms of severe pulmonary dysfunction. PFT testing must show FEV1 and DLCOcorr > 50% of predicted if subjects have symptomatic or prior known impairment.
  * Transthoracic echocardiogram with PA pressures in the range of 18-26 mmHg
  * Ability to be off prednisone and other immunosuppressive drugs for at least 14 days before infusion of cells
  * Women of child bearing potential and men with partners of child bearing potential must agree to use effective contraception during therapy and for 4 months after completion of therapy
  * Voluntary written consent provided by the subject

Exclusion Criteria:

* Any condition that precludes lymph node biopsy or colonoscopy with biopsy

  * Active infection other than HIV currently requiring systemic antimicrobial therapy
  * History of deep vein thrombosis
  * Active significant, tissue invasive fungal infection requiring systemic antifungal therapy (dermatologic conditions requiring only topical therapy are allowed).
  * Chronic active hepatitis B or C (defined as antibody positive and DNA+ or HepBsAG+).
  * Breastfeeding
  * Intended modification of antiretroviral therapy in the next 24 weeks
  * NYHA (New York Heart Association) Class III or IV heart failure, uncontrollable supraventricular arrhythmias, any history of a ventricular arrhythmia, or other clinical signs of severe cardiac dysfunction
  * Symptomatic congestive heart failure, unstable angina pectoris, or Myocardial infarction within 6 months prior to screening
  * Marked baseline prolongation of QT/QTc interval (e.g. demonstration of a QTc interval greater than 500 milliseconds)
  * On-going chronic systemic corticosteroid use or other immunosuppressive therapy (a history of mild asthma not requiring therapy is eligible and inhaled corticosteroids is allowed. Topical steroids are allowed.)
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Previous diagnosis of an autoimmune disease (e.g. rheumatoid arthritis, lupus, inflammatory bowel disease, multiple sclerosis, vasculitis)
  * Use of any anticoagulants within the previous 4 weeks.
  * Other illness that in the opinion of the investigator would exclude the patient from participating in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Safety of administration of haploidentical NK cells in HIV infected individuals - Adverse Events | Baseline, 100 days
  Subjects will receive haploidentical NK and all adverse events will be collected
Tolerability of administration of haploidentical NK cells in HIV infected individuals- Side effects | Baseline, 100 days
  Side effects from all subjects will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Schacker, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Miller JS, Rhein J, Davis ZB, Cooley S, McKenna D, Anderson J, Escandon K, Wieking G, Reichel J, Thorkelson A, Jorstad S, Safrit JT, Soon-Shiong P, Beilman GJ, Chipman JG, Schacker TW. Safety and Virologic Impact of Haploidentical NK Cells Plus Interleukin 2 or N-803 in HIV Infection. J Infect Dis. 2024 May 15;229(5):1256-1265. doi: 10.1093/infdis/jiad578. PMID 38207119